CLINICAL TRIAL: NCT05654493
Title: Use of Micropulse Trans-Scleral Cyclophotocoagulation Laser (MP-TSCPC) for Glaucoma Patients: Clinical Outcomes. Prospective Observational Cohort Study
Brief Title: Use of Micropulse Trans-Scleral Cyclophotocoagulation Laser (MP-TSCPC) for Glaucoma Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Syril K. Dorairaj, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-008815
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- 240 Second Group (Experimental): Receives 240 seconds total of MicroPulse Transscleral Laser Therapy with the revised P3 Delivery Device delivered in a total of 8 sweeps
  Interventions: Device: MicroPulse Transscleral Laser Therapy using revised P3 Delivery Device
- 300 Second Group (Experimental): Receives 300 seconds total of MicroPulse Transscleral Laser Therapy with the revised P3 Delivery Device delivered in a total of 10 sweeps
  Interventions: Device: MicroPulse Transscleral Laser Therapy using revised P3 Delivery Device
- 200 Second Group (Experimental): Receives 200 seconds total of MicroPulse Transscleral Laser Therapy with the revised P3 Delivery Device delivered in a total of 8 sweeps
  Interventions: Device: MicroPulse Transscleral Laser Therapy using revised P3 Delivery Device

INTERVENTIONS:
Device: MicroPulse Transscleral Laser Therapy using revised P3 Delivery Device — The MicroPulse G-Probe was applied to the superior and inferior hemispheres of the eye under varied treatment times and sweep numbers
  Other Names: MP-TLT

SUMMARY:
The purpose of this study is to evaluate the clinical outcomes of the Micropulse Trans-Scleral Cyclophotocoagulation Laser (MP-TSCPC) after 1 day, 1 week,1 month, 3 months, 6 months and one year of follow-up, with the intent to evaluate the efficacy of using MP-TSCPC to treat glaucoma patients.

DETAILED DESCRIPTION:
Patients will be submitted to MP-TSCPC throughout the year of 2020, according to parameters determined by the Principal Investigator and executed by the Principal Investigator, after signing the Consent Form and agreeing on having their data used for research purpose. Postsurgical follow up visits will be scheduled for 1 month, 3 months, 6 months and 12 months. Patients IOP, number of medications, visual acuity, visual field, iris color, retinal nerve fiber layer thickness on OCT and any complications (iritis, corneal edema, hyphema, vitreous hemorrhage, vision loss, cataract progression or hypotony maculopathy) will be measured by trained ophthalmic assistants supervised by the Principal Investigator and documented at each visit. Authorized Mayo Clinic personnel will perform chart reviews; using administrative data as designated by Dr. Dorairaj. The data will be statistically analyzed to illustrate the results and determine if the objectives and primary and secondary endpoints were achieved

ELIGIBILITY:
Inclusion Criteria:

* Diagnose of glaucoma
* Indication to be submitted to the procedure

Exclusion Criteria:

* Significant thinning of the sclera
* Current eye infection or inflammation
* Intraocular surgery performed less than 2 months prior to the enrollment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change In IOP | Baseline, 12 months post procedure
  Change in intraocular pressure (IOP), reported in millimeters of mercury (mm Hg)

SECONDARY OUTCOMES:
Number of anti-glaucoma medications | 12 months
  Number of anti-glaucoma medication drops
Change in visual acuity | Baseline, 12 months post procedure
  Change in visual acuity score
Change in cup-disc ratio | Baseline, 12 months post procedure
  Ratio of the size of the optic cup to the optic disc
Change in visual field | Baseline, 12 months post procedure
  Total area visible in peripheral vision when focused on a central point, reported in degrees
Change in iris color | Baseline, 12 months post procedure
  Number of subjects to have a change in their iris color
Complications | 12 months
  Number of subjects to experience complications from the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Syril Dorairaj, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20477448